CLINICAL TRIAL: NCT05958940
Title: BioClock: Optimization, Working Mechanisms and Response Predictors of Bright Light Therapy for Depressive Disorders - a Multicentre Randomized Controlled Trial
Brief Title: BioClock: Bright Light Therapy for Depressive Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Leiden (Other)
Collaborators: Eindhoven University of Technology (Other); Geestelijke Gezondheidszorg Eindhoven (GGzE) (Other); Chrono@Work B.V. (Unknown)
Responsible Party: Principal Investigator, Niki Antypa, Associate Professor, Universiteit Leiden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL83497.058.23
Record Dates: First submitted 2023-07-07; First posted 2023-07-25 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Depression, Unipolar; Depression, Bipolar
Keywords: Depression; Bright Light Therapy; Chronotherapy; Circadian Rhythm; Sleep; Life Style; Ecological Momentary Assessment; Actigraphy; Dim light melatonin onset; Response predictors
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder; Depression | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Light@Home (Active Comparator): Standard Care - BLT in the home environment
  Interventions: Procedure: Bright Light Therapy
- LightCafé (Experimental): BLT will be administered in a specialized cafe, under the supervision of clinical staff, promoting lifestyle changes and social interaction.
  Interventions: Procedure: Bright Light Therapy
- LightCafé+ (Experimental): Treatment will be identical to the second arm but now complemented with the use of blue-light blocking glasses in the evening and the adoption of personalized BLT timing based on sleep-wake patterns
  Interventions: Procedure: Bright Light Therapy; Device: Blue Light Blocking Glasses

INTERVENTIONS:
Procedure: Bright Light Therapy — In this study, Bright Light Therapy (BLT) will be administered according to Dutch depression guidelines, using Innolux LED light lamp (3800K, 10,000 lux). BLT will be given for one work week (Mon-Fri), 7:30-10:30 AM, 30 mins/session. Patients can have breakfast, read, or use devices. Treatment effectiveness will be evaluated using Self-Rated Quick Inventory of Depressive Symptoms (QIDS-SR). If remission is achieved (QIDS-SR < 6), no additional treatment is given. If response is insufficient (QIDS-SR ≥ 6), 5 more sessions will be added in the following week, with maximum two extensions (1-3 weeks total).
Device: Blue Light Blocking Glasses — Plastic, orange-coloured glasses that primarily block blue light. To be worn in the evening.
  Arms: LightCafé+

SUMMARY:
Bright Light Therapy (BLT) is a proven treatment for depression in seasonal and non-seasonal depressive disorders, as well as bipolar disorder. To make BLT more effective and practical in clinical settings and tailor it to individual needs, it is necessary to optimize the treatment approach, understand how the treatment works, and identify patient characteristics that predict response.

This clinical trial has three main goals:

* Optimize the administration of BLT for patients with depressive episodes.
* Gain a deeper understanding of the treatment mechanisms.
* Determine which patients benefit the most from the treatment.

The specific objectives are as follows:

* Investigate whether additional treatments and interventions related to lifestyle and the biological clock can enhance the effects of BLT.
* Examine how BLT influences the body's internal clock and sleep quality, and how these factors contribute to the outcomes.
* Identify patient characteristics and behaviours that can predict treatment outcomes.
* Develop a brain model to better understand the impact of BLT on the brain.

In this study, patients will receive BLT with a light intensity of 10,000 lux for 30 minutes each morning over 5 consecutive days. The treatment duration will range from one to three weeks, depending on the improvement of depressive symptoms. Participants will be randomly assigned to one of three groups:

* Home - Patients will receive BLT at home, following the standard guidelines for light therapy in the Netherlands.
* LightCafé, fixed time: Patients will receive BLT in a café-like setting called the LightCafé, where the focus is not only on symptom improvement but also lifestyle enhancements and fostering social connections. The treatment time will be the same every day.
* LightCafé, varying time: Patients will also receive BLT at the LightCafé, with treatment timing varying each day. Additionally, this group will wear glasses in the evening that filter blue light.

The study includes a baseline phase of up to two weeks, a treatment phase of up to three weeks, and a three-month follow-up phase. Patients will wear a motion watch to assess sleep-wake behaviour and physical activity during the day. Additionally, they will wear a broach that measures their personal light exposure throughout the day. Eight one-minute questionnaires per day will be sent to the participants' smartphones to assess vitality, sleep, and mood during the treatment. Predictors of treatment response, such as clinical characteristics, sleep measures, circadian parameters, and light-related behaviours, will be evaluated at baseline. In a small group of patients, salivary melatonin curves will be assessed before and after treatment. MRI scans will provide insights into functional and structural brain changes following light therapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65.
* Diagnosis of unipolar or bipolar depression (seasonal or non-seasonal) as assessed with the Mini-International Neuropsychiatric Interview (M.I.N.I.)
* A current depressive episode (a score of 6 or higher on the Quick Inventory of depressive symptomatology Self Report (QIDS-SR)
* Sufficient knowledge of Dutch or English language to fill in questionnaires
* Provided Informed consent

Exclusion Criteria:

* A current (hypo)manic or mixed episode (as assessed with the M.I.N.I.)
* Current psychotic episode (as assessed with the M.I.N.I.)
* Prominent active suicidality (score 10 or higher on the M.I.N.I. module)
* Antidepressant therapy (medication, psychotherapy or BLT, or other forms of specific treatments for depression) that started less than 2 months prior to study entry
* participants with bipolar disorder should be in mood-stabilizing treatment for at least 1 month in a recommended dosage,
* Use of melatonin or agomelatine in the last month
* Current use of antibiotics
* Current use of light sensitivity increasing medication
* Travelled across more than 1 time zone during past month or during the treatment
* Travelled to sunny holiday locations/winter sports during past month
* pre-existing eye and skin disorders (retinitis pigmentosa, porphyria, chronic actinic dermatitis and sun-induced urticaria)
* Systemic disorders with potential retinal involvement (rheumatoid arthritis and systemic lupus erythematosus)
* Suffering from colour blindness (assessed by Ishihara colour plates)
* Participated in night shift work in the last three months
* (Retinal) blindness, severe cataract and glaucoma
* Light-induced migraine or epilepsy
* Pregnancy, or parents with a child younger than 18 months old

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Improvement | 2-5 weeks
  Difference between pre- and post-treatment assessment of the Montgomery Asberg Depression Rating Scale [MADRS]

SECONDARY OUTCOMES:
Subjective change in depressive symptom severity | from baseline until follow-up, approximately 4 months
  Change in score on the Quick Inventory of Depressive Symptoms, Self Report (QIDS-SR)
Remission rates, self assessed and clinician rated | 2-5 weeks for clinician rated. Up until 4 months after start treatment for self-assessed
  percentage of patients that after treatment have a score of <6 on the MADRS or QIDS-SR
Response Rates, self assessed and clinician rated | 2-5 weeks for clinician rated, Up until 4 months after start treatment for self-assessed
  percentage of patients hat after treatment have at least 50% reduction in depressive symptom, measured using MADRS and QIDS-SR
Time to remission | one, two or three weeks
  The time it takes to achieve remission, if remission is achieved. Measured with QIDS-SR
Circadian phase | 2-5 weeks
  Changes in circadian phase will be compared between groups as assessed using the DLMO (calculated from the melatonin assessments) and complemented with actigraphy data (using sleep onset timing, least active 5h period and most active 10h period)
Circadian amplitude | 2-5 weeks
  Changes in the circadian amplitude will be compared between groups. The amplitude can be estimated from actigraphy data by the difference in activity between the most active 10h and the least active 5h normalized for total activity.
Circadian Periodicity | 2-5 weeks
  Changes in circadian periodicity will be compared between groups. Circadian periodicity is a period of an oscillating rhythm assessed via periodogram analysis of the activity time-course of actigraphy data. The deviation between the maximum period of the periodogram and the normal daily period of 24h reflects pattern variability in normal entrainment conditions.
Inter-daily stability | 2-5 weeks
  Constancy of the 24-h rhythmic pattern over days
Intra-daily variability | 2-5 weeks
  rhythm fragmentation
Chronotype | 1-3 months
  Chronotype changes as assessed with the Morningness-Eveningness Questionnaire(MEQ) and the Ultra-Short Version of the Munich Chronotype Questionnaire (µMCTQ)
Sleep-Wake Pattern | 2-5 weeks
  Actigraphy and questions from The Consensus Sleep Diary will provide sleep onset time, sleep offset time, midsleep time, total sleep time, sleep onset latency, number of awakenings and time awake during the night.
Sleep Quality | 2-5 weeks for actigraphy, up until 4 months after the start of treatment for subjective sleep quality
  Fragmentation index (degree of movement during the night), sleep efficiency (total sleep time expressed as a percentage of time in bed) will be calculated using actigraphy data. The Pittsburgh Sleep Quality Index (PSQI) will provide a subjective measure of sleep quality.
Severity of Insomnia Symptoms | up until 4 months after the starts of treatment
  Severity of Insomnia Symptoms as assessed with the Insomnia Severity Index
Momentary Positive/Negative Affect | 2-5 weeks
  The EMA will consist of items from the Positive and Negative Affect Scale (PANAS) to assess momentary positive and negative affect
Momentary Vitality | 2-5 weeks
  The EMA will contain 4 items concerning energy levels and alertness adapted from Activation-Deactivation Adjective Checklist
Gray matter structure | 2-5 weeks
  Properties of gray matter structure (thickness, volume, surface area and gyrification) of the whole brain as well as of the white matter structure (integrity of main white matter fiber tracts-fractional anisotropy (FA))
Functional connectivity of the brain | 2-5 weeks
  Functional connectivity of the brain under resting state condition - the communication of specific brain regions which work as a network without conducting a specific task

OTHER OUTCOMES:
Personal daily light exposure | 2-5 weeks
  the percentage of time exposed to light above the threshold of 300 lux will be calculated from light sensor data as well as the mean timing thereof (MLiT100). Additional parameter might be extracted from the light exposure data based on state of the art procedures.
Treatment expectations | baseline
  Treatment expectations will be assessed using the Credibility/expectancy Questionnaire
Light Induced Melatonin suppression | Baseline
  Light Induced Melatonin suppression as assessed using the salivary melatonin assessments will give insight into light sensitivity of the participants.
Treatment Adherence | 1-3 weeks
  Treatment adherence will be assessed subjectively using an item in the EMA and objectively using light logger devices.
Side Effects | 1-3 weeks
  Side effects will be monitored with a questionnaire based on the Toronto Side Effects Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Niki Antypa, PhD, Principal Investigator — Leiden University
Locations (2):
- Netherlands (2):
  - GGzE - Mental Health Institute of Eindhoven and the Kempen, Eindhoven
  - Leids Universitair Behandel- en Expertise Centrum, Leiden

IPD SHARING:
Plan to Share IPD: Yes
All data underlying a publication can be shared upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after publication of the analyses
Access Criteria: Access may be granted to researchers who intend to conduct secondary analyses or meta-analyses using individual participant data. Additionally, researchers with a valid scientific research question or hypothesis that aligns with the objectives of the original study may be considered for IPD access.

REFERENCES:
- [Derived] Visser E, Rus-Oswald OG, van der Does AJW, Gordijn MCM, Marcelis MC, de Kort YAW, Oomen PP, Schlangen LJM, Seetsen T, Simons CJP, Antypa N. BioClock-optimizing Bright Light Therapy for adults with depression: a study protocol for a multicenter randomized clinical trial on treatment strategies, response predictors, and chronobiological and neurobiological mechanisms. Trials. 2025 Oct 14;26(1):411. doi: 10.1186/s13063-025-08984-7. PMID 41088238